CLINICAL TRIAL: NCT05443646
Title: A Phase II Study of Consolidation HLX10 (Serplulimab) Following Hypofractionated Radiotherapy With Concurrent Chemotherapy for Patients With Limited Stage Small Cell Lung Cancer
Brief Title: Consolidation Serplulimab Following Concurrent Chemoradiotherapy for LS-SCLC Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ASTRUM-LC01
Record Dates: First submitted 2022-06-29; First posted 2022-07-05 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Limited Stage Small Cell Lung Cancer
MeSH Terms: interventions — Radiation Dose Hypofractionation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HLX10 (Serplulimab) Consolidation After Chemotherapy Concurrent Hypofractionated Radiotherapy (Experimental): Participants will receive at least 4 cycles of standard-of-care chemotherapy (carboplatin/cisplatin-etoposide) concurrently with Hypofractionated Radiotherapy, followed by HLX10 300 mg every 3 weeks (Q3W) with maximum 1 years or until disease progression, intolerable toxicity or other reasons specified in the protocol, whichever occurs first.
  Interventions: Drug: HLX10; Radiation: hypofractionated radiotherapy; Radiation: Prophylactic Cranial Irradiation (PCI)

INTERVENTIONS:
Drug: HLX10 — HLX10 is an innovative monoclonal antibody targeting PD-1，developed by Shanghai Henlius Biotech, Inc.
  300mg Q3W
  Other Names: Serplulimab
Radiation: hypofractionated radiotherapy — 45Gy/3Gy/3week
Radiation: Prophylactic Cranial Irradiation (PCI) — 25Gy/2.5Gy/2week

SUMMARY:
This study is a multi-center, Single-arm Phase II study to evaluate the clinical efficacy and safety of Consolidation HLX10 (Serplulimab) Following Hypofractionated Radiotherapy With Concurrent Chemotherapy for Patients With Limited Stage Small Cell Lung Cancer

DETAILED DESCRIPTION:
All eligible patients after screening will receive up to four cycles chemotherapy. Recommended regimens are etoposide 100 mg/m2 intravenously on day 1-3 in combination with cisplatin 75 mg/m2 intravenously on day 1 or carboplatin AUC=5 every 3 weeks.

A total of 45Gy in 15 fractions over 3 weeks will be delivered. PCI is routinely scheduled for patients without progression after chemoradiotherapy, and hippocampal avoidance is highly recommended. 25Gy in 10 fractions over 2 weeks to the brain will be prescribed. Intensity modulated radiation therapy (IMRT) or volumetric modulated arc therapy (VMAT) technique are required. Patients without disease progression will receive an intravenous infusion of serplulimab 300mg every 3 weeks. Treatment of serplulimab should be continued until disease progression, intolerable toxicity, withdrawal of consent, or to a maximum of 1 year. Continuation of immunotherapy after disease progression is acceptable per investigators' discretion.

The investigator and IRRC respectively assess the tumor images according to RECIST 1.1.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years; ECOG score 0-1.
2. Histologically or cytologically confirmed small cell lung cancer.
3. Limited stage, defined as the tumor confined to one side of the thoracic cavity including ipsilateral hilar, bilateral mediastinal, and bilateral supraclavicular lymph nodes, (metastatic lymph nodes are defined as short diameter ≥ 1 cm or increased metabolism on PET-CT considering metastatic lymph nodes); unless cytologically confirmed malignant pleural effusion, the thickness of pleural effusion on chest CT is less than 1 cm; (stage I-IIIB without intrapulmonary metastasis in the 7th edition of AJCC staging in 2009) .
4. No other previous anti-tumor history, at least 3 months of expected survival.
5. No serious medical diseases and dysfunction of major organs, such as blood routine, liver, kidney, heart and lung function.

Exclusion Criteria:

1. Histologically or cytologically confirmed mixed SCLC.
2. Subjects suitable for surgery. Subjects who are suitable for surgery but refuse surgical treatment can be included.
3. Patients who have previously received systematic anti-tumor treatments for small cell lung cancer, including but not limited to radiotherapy, chemotherapy, and immunotherapy.
4. Patients with other active malignancies within 5 years or at the same time.
5. Subjects with known history of severe allergy to any monoclonal antibody.
6. Subjects with known anaphylaxis to carboplatin/cisplatin or etoposide.
7. In the judgment of the investigator, subjects who have any other factors that may lead to a premature discontinuation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2022-09-23 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | up to 12 months
  To evaluate the progression-free survival (PFS) of HLX10 (Serplulimab) consolidation therapy after concurrent hypofractionated radiotherapy with chemotherapy in limited-stage small cell lung cancer according to RECIST 1.1 criteria

SECONDARY OUTCOMES:
Overall survival(OS） | up to 24 months
  Overall survival time is defined as the time from the date of the patient's first dose of HLX10 to the date of any documented death due to any cause.
Objective response rate (ORR) | up to 24 months
  Proportion of subjects achieving a best response of complete response (CR) and partial response (PR) as assessed by RECIST 1.1.
Time to treatment failure (TTF) | up to 12 months
  Time to disease progression, death, withdrawal due to adverse events, patient refusal to continue the study, or use of a new treatment from the first HLX10 administration.

CONTACTS AND LOCATIONS:
Overall Officials: Nan Bi, Doctor, Principal Investigator — Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College
Locations (2):
- China (2):
  - Jiamusi Cancer Hospital, Jiamusi, Heilongjiang
  - Shanxi Province Cancer Hospital, Taiyuan, Shanxi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wu Y, Deng L, Wang J, Zhang T, Cao J, Zhou X, Duan J, Bi N. Single-arm phase II study of consolidation serplulimab following hypofractionated radiotherapy with concurrent chemotherapy for patients with limited stage small-cell lung cancer: ASTRUM-LC01 study protocol. BMJ Open. 2025 May 21;15(5):e085552. doi: 10.1136/bmjopen-2024-085552. PMID 40398957